CLINICAL TRIAL: NCT07194044
Title: Metastatic Ewing's Trial Testing Schedule Enhancement to Improve Outcomes
Acronym: METTSEO
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: National Pediatric Cancer Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-23281
Record Dates: First submitted 2025-09-17; First posted 2025-09-26 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Metastatic Ewing Sarcoma
MeSH Terms: conditions — Sarcoma, Ewing | interventions — Vincristine; Doxorubicin; Cyclophosphamide; Ifosfamide; Dactinomycin; Irinotecan; cabozantinib; Topotecan; Temozolomide; Etoposide; liposomal doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Sequential Therapy (Experimental): Weeks 1-8, Vincristine/Doxorubicin/Cyclophosphamide. Weeks 9-14, Irinotecan, Ifosfamide, Vincristine, Actinomycin (IrIVA). Weeks 15-20, Cabozantinib w/ primary site radiation. Weeks 21-26, Topotecan/Cyclophosphamide. Weeks 27-32, High Dose Ifosfamide. Weeks 33-38, Irinotecan/Temozolomide. Maintenance, Weeks 39 up to 104, will consist of alternating 28-day blocks of chemotherapy (Block 1 and Block 2). Oral Cyclophosphamide / Oral Etoposide (Block 1). Vincristine/ Liposomal Doxorubicin (Block 2).
  Interventions: Drug: Vincristine; Drug: Doxorubicin; Drug: Cyclophosphamide; Drug: Ifosfamide; Drug: Actinomycin; Drug: Irinotecan; Drug: Cabozantinib; Drug: Topotecan; Drug: Temozolomide; Drug: Etoposide; Drug: Liposomal doxorubicin

INTERVENTIONS:
Drug: Vincristine — IV Push
Drug: Doxorubicin — IV
Drug: Cyclophosphamide — IV and Maintenance PO
Drug: Ifosfamide — IV
Drug: Actinomycin — IV
Drug: Irinotecan — IV
Drug: Cabozantinib — PO
Drug: Topotecan — IV
Drug: Temozolomide — IV
Drug: Etoposide — PO
Drug: Liposomal doxorubicin — IV

SUMMARY:
This single arm study is designed to demonstrate the feasibility of a radically different approach for an exceptionally high-risk subset of MES with widely metastatic disease (WMES). We incorporate the use of evolutionary principles that apply to species and population dynamics as related to adaptation and extinction to populations of cancer cells that similarly adapt and that we are attempting to make extinct, resulting in a cure for the patient. Such principles include an initial intense first strike to deplete the bulk of the cancer cells, followed by a series of sequential second strikes towards eliminating residual, resistant populations, followed by a prolonged period of maintenance chemotherapy to eliminate any remnant cells, using agents generally regarded to be active against newly diagnosed ES.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be >1 year of age. There is no upper age limit.
* Patients, in the opinion of the enrolling investigator, must be healthy enough to tolerate protocol therapy.
* Patients must have a new histologic diagnosis of either: widely metastatic Ewing sarcoma or metastatic CIC-rearranged sarcoma.
* Patients must have sufficient tissue submitted (flash frozen tissue, FFPE block, or up to 10 unstained FFPE slides) for correlative testing. This may be from a primary or metastatic site.
* Patients must not have received any prior systemic therapy with the exception that they may have started an initial cycle of vincristine/doxorubicin/cyclophosphamide (VDC) prior to enrollment, i.e. VDC may have been given, but not ifosfamide/etoposide (IE).
* Adequate organ function.
* Males and females of reproductive potential may not participate unless they have agreed to the use of, at minimum, two methods of contraception during and after treatment or abstinence.
* All patients and/or their parents or legal guardians must have the ability to understand and the willingness to sign a written informed consent or assent document.

Exclusion Criteria:

* Patients with localized disease or lung only metastases for Ewing sarcoma or localized disease for CIC-rearranged sarcomas.
* Patients with central nervous system (CNS) tumors (primary or metastatic) are not eligible.
* Patients who are receiving any other investigational agents for their cancer.
* Patients with a history of cancer that was treated with myelosuppressive chemotherapy or radiation therapy.
* Patients must not be receiving any additional medicines being given for the specific purpose of treating cancer.
* Patients are ineligible if they have uncontrolled intercurrent illness.
* Pregnancy or Breast Feeding: Pregnant or breast-feeding women will not be entered on this study, because there is no available information regarding human fetal or teratogenic toxicities. Females of childbearing potential must have a negative serum or urine pregnancy test within 72 hours prior to starting protocol therapy.
* Patients who are considered unable to comply with the safety monitoring requirements of the study are not eligible.

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2030-10 (Estimated); Study Completion 2030-10 (Estimated)

PRIMARY OUTCOMES:
Feasibility and Safety - Consolidation | 16 months
  The treatment will be considered feasible if 70% of Ewing sarcoma patients make it through consolidation.
Feasibility and Safety - Maintenance | 16 months
  The treatment will be considered feasible if 50% of Ewing sarcoma patients make it through 6 cycles of maintenance.

SECONDARY OUTCOMES:
Event-Free Survival | 3 years
  EFS is defined as time from treatment initiation to event which includes (1) recurrence, (2) secondary malignancy, and (3) death due to any cause.
Off Treatment Event Free Survival | 3 years
  otEFS is defined as time from treatment initiation to event 66 which includes (1) any recurrence (local or regional, or distant) that leads to coming off protocol therapy and (2) death due to any cause.
Overall Survival | 3 years
  The time to event endpoint of overall survival is defined as the duration of time from diagnosis to death or last follow-up timepoint, where event would be death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Matteo Trucco, MD, Principal Investigator — Cleveland Clinic Hospital; Jonathan Metts, MD, Principal Investigator — Moffitt Cancer Center
Locations (17):
- United States (17):
  - University of Alabama at Birmingham (Children's of Alabama), Birmingham, Alabama
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - University of Florida, Gainesville, Florida
  - Nemours Jacksonville, Jacksonville, Florida
  - University of Miami, Miami, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - University of Kentucky, Lexington, Kentucky
  - Helen DeVos Children's Hospital, Grand Rapids, Michigan
  - Roswell Park Comprehensive Cancer Center, Buffalo, New York
  - Montefiore Medical Center, The Bronx, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Levine Cancer Institute, Charlotte, North Carolina
  - Cleveland Clinic Children's, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Primary Children's Hospital, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Undecided